CLINICAL TRIAL: NCT06160869
Title: Efficacy of Acceptance and Commitment Therapy on Psychotic Severity Among Inpatients With Primary Psychosis: A Randomized Controlled Trial.
Brief Title: Effect of Acceptance and Commitment Therapy on Psychotic Severity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Port Said University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P.0553
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-10

CONDITIONS: Psychosis; Emotion Regulation; Recovery
Keywords: Psychosis; Emotional regulation; Recovery
MeSH Terms: conditions — Psychotic Disorders; Emotional Regulation | interventions — Acceptance and Commitment Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Current study is an open label, two-arm, parallel, randomized controlled trial, evaluating the efficiency of Acceptance and Commitment Therapy (ACT) added to treatment as usual (TAU) as opposed to treatment as usual (TAU) alone on patients with schizophrenia. The study adheres to the rules for writing Clinical Trials: "The Consolidated Standards of Reporting Trials" (CONSORT) statement
Masking Description: Information is not withheld from trial participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT Group (Experimental): Received 90-minutes weekly group sessions of acceptence and commitment therapy plus treatment as usual.
  Interventions: Behavioral: Acceptance and commitment therapy
- Treatment as usual (TAU) group (Active Comparator): Will receive the TAU alone
  Interventions: Combination Product: Treatment as usual

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — The psychoeducational intervention will consist of seven structured sessions aimed at introducing patients with primary psychosis to the principles and practices of Acceptance and Commitment Therapy (ACT). The primary focus of the intervention is to empower participants to effectively manage distressing thoughts and feelings while pursuing meaningful and valued life goals. Each session covers specific aspects of ACT.
  Acceptance and commitment therapy will be adminitered in addition to treament as usual provided to patients.
  Arms: ACT Group
Combination Product: Treatment as usual — The treatment as usual (TAU) for all patients regardless of condition will consist of hospital treatment, including daily medication management sessions with a psychiatrist (e.g., antipsychotic and other medications as appropriate), community meetings, other group therapy, case management, occupational therapy, open air walks, discharge planning, physical examination, and other services (e.g., medical testing).
  Arms: Treatment as usual (TAU) group

SUMMARY:
Our study aims to assess the efficacy of Acceptance and Commitment Therapy on psychotic severity among Inpatients with primary psychosis: A Randomized Controlled Trial.

DETAILED DESCRIPTION:
Current study was an open label, two-arm, parallel, randomized controlled trial, evaluating the efficiency of Acceptance and Commitment Therapy (ACT) added to treatment as usual (TAU) as opposed to treatment as usual (TAU) alone on patients with schizophrenia. The study adheres to the rules for writing Clinical Trials: "The Consolidated Standards of Reporting Trials" (CONSORT) statement

ELIGIBILITY:
Inclusion criteria Participants' criteria of inclusion involved those patients who were

1. Current psychiatric hospitalization;
2. DSM-5 diagnosis of a primary psychotic disorder; (schizophrenia, schizoaffective disorder, delusional disorder, schizophreniform disorder, brief psychotic disorder, and unspeciﬁed psychotic disorder, this diagnosis was confirmed by a psychiatrist
3. 18 years or older;
4. ability to talk, read and write in Arabic; and
5. willingness to participate in the study that was scheduled for seven weeks.

Exclusion criteria Patients were excluded if they

1. had a comorbid learning disability or organic brain disorder;
2. psychosis related to a general medical condition or substance-induced psychotic disorder;
3. were considered mentally unstable; or
4. unfit to participate in the study by their therapist, and/or had newly had (been receiving) psycho-education or somewhat designed psychosocial intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 7 weeks
  Measuring symptom severity of patients with schizophrenia. This is a 30-item instrument. Rating of each item is from (one, no evidence) to (seven, strong evidence) and the total score for overall psychopathology ranges from 30 to 210.

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale | 7 weeks
  A 36 item measure assesses individuals' typical levels of difficulties in emotion regulation
Recovery Assessment Scale | 7 weeks
  38 items scale evaluate mental health recovery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Zoromba, PhD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
To ensure privacy and confidentiality of participants their data will be secured

REFERENCES:
- [Derived] Zoromba MA, Sefouhi L, Alenezi A, Selim A, Awad S, El-Gazar HE, El-Monshed AH. Effectiveness of Acceptance and Commitment Therapy on Psychotic Severity Among Inpatients With Primary Psychoses: A Randomized Controlled Trial. Int J Ment Health Nurs. 2024 Dec;33(6):2239-2256. doi: 10.1111/inm.13388. Epub 2024 Jul 21. PMID 39034443